CLINICAL TRIAL: NCT04092257
Title: A Novel Cervical Cancer Screen-and-Treat Demonstration Project With HPV Self-testing and Thermocoagulation for Women in Lilongwe Malawi
Brief Title: HPV-Based Screen-and-Treat Demonstration Project in Lilongwe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1905; R21CA236770 (NIH); AID-OAA-A-11-00012 (Other Grant/Funding Number: USAID/NAS)
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: HPV Infection; Cervical Cancer; HIV Infections
Keywords: Visual inspection with acetic acid (VIA)
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; HIV Infections | interventions — Electrocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIA and thermocoagulation (Experimental): Participants will undergo same day VIA and thermocoagulation
  Interventions: Procedure: VIA and thermocoagulation

INTERVENTIONS:
Procedure: VIA and thermocoagulation — Participants will self-collect a vaginal brush for hr-HPV testing. HPV-positive women and every 10th consecutive HPV-negative woman will complete same-day VIA with colposcopically-directed cervical biopsy and ECC (if lesion seen), and thermocoagulation if ablation-eligible by colposcopy. If no lesion is seen on colposcopy, the woman will have a cervical pap smear and ECC collected, and no thermocoagulation will be performed. Finally, women who are suspicious for cancer at VIA will undergo colposcopically-directed cervical biopsies.

SUMMARY:
The purpose of this study is to assess completion and performance of the following novel invasive cervical cancer (ICC) screen-and-treat algorithm among 625 HIV-positive women in Lilongwe, Malawi: 1) rapid testing of self-collected vaginal brush for primary high risk (hr)-human papillomavirus (HPV), 2) same-day visual inspection with acetic acid (VIA) for women who are hr-HPV positive, and 3) thermocoagulation for VIA positive/ablation-eligible (by cervical colposcopy) women.

DETAILED DESCRIPTION:
This is a single arm, prospective study of 1,250 women (625 HIV-positive and 625 HIV-negative) enrolled from outpatient clinics that provide sexual and reproductive health (SRH) services and/or HIV care services in Lilongwe, Malawi. The primary objectives of this study are to assess completion of a novel ICC screen-and-treat strategy among HIV-positive women in Lilongwe, Malawi, using self-collected vaginal brush for hr-HPV testing, followed by same-day NIA and thermocoagulation for HPV-positive/NIA-positive/ablation-eligible (by colposcopy) women, and to determine the 24-week efficacy of thermocoagulation among HIV-positive women with CIN2/3. The secondary objective will be to evaluate the performance of the ICC screen-and-treat strategy by estimating overtreatment for women who are HPV-positive/NIA-positive/ablation-eligible, and undertreatment among HPV-positive/NIA-negative women.

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥ 25 years of age at study entry and ≤ 50 years of age (per current Malawi National Cervical Cancer Control Program guidelines for screening).
2. Ability and willingness of participant to provide written informed consent.

Exclusion Criteria:

1. Current or prior history of cervical, vaginal, or vulvar cancer or dysplasia
2. Current symptomatic sexually transmitted infection requiring treatment (women will be allowed to be in the study upon successful treatment)
3. Prior HPV vaccination.
4. Participants with known allergy to acetic acid.
5. Participants with a history of total hysterectomy.
6. Participants who are pregnant or plan on becoming pregnant during the study period.
7. Participants who are less than 12 weeks postpartum.
8. Participants with other illnesses that would limit compliance with study requirements or in the opinion of the investigator or designee, have a problem that would make participation in the study unsafe or complicate interpretation of study findings.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1250 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lameck Chinula, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina (UNC) Project-Malawi, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from health facilities with outpatient clinics that provide sexual and reproductive health services and/or HIV care services in Lilongwe, Malawi between 6/24/2020- 2/28/2022. The first participant was enrolled on 6/24/2020, and the last participant was enrolled on 2/28/2022.
Pre-assignment Details: Participants were assigned HIV-positive or HIV-negative groups based on HIV testing result.
Groups:
- HIV Positive: Women living with HIV
- HIV Negative: Women living without HIV
Period: Overall Study
Arm/Group | HIV Positive | HIV Negative
Started | 625 | 625
Completed | 602 | 618
Not Completed | 23 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Positive | HIV Negative | Total
Number analyzed (Participants) | 625 | 625 | 1250
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [33 to 41] | 33 [28 to 38] | 35 [30 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 625 | 625 | 1250
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 625 | 625 | 1250
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 625 | 625 | 1250
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 625 | 625 | 1250
Level of education [Count of Participants; unit: Participants]
  No education | 94 | 39 | 133
  Primary | 344 | 305 | 649
  Secondary | 172 | 245 | 417
  Tertiary | 15 | 36 | 51
Marital status [Count of Participants; unit: Participants]
  Never married | 9 | 29 | 38
  Married/Living with partner | 395 | 475 | 870
  Widowed/divorced/separated | 221 | 121 | 342

OUTCOME MEASURES:

1. Primary Outcome: Same-day Visual Inspection With Acetic Acid (VIA) Rate
Description: The proportion of women who were HPV-positive and underwent same-day VIA following self-collected vaginal sampling was assessed, including both HIV-positive and HIV-negative participants. As per the study protocol, data were not stratified by HIV status for this outcome due to lack of scientific rationale for a difference in same-day VIA completion by HIV status.
Time Frame: Baseline
Population: Participants who underwent HPV-based primary screening for cervical cancer and tested HPV-positive on self-collected vaginal sample and had VIA triage performed on the same day of self-collection.
Measure: Count of Participants; unit: Participants
Groups:
- HPV Positive: All HPV positive women.
Arm/Group | HPV Positive
Number analyzed (Participants) | 476
Participants
  Visual Inspection with Acetic Acid (VIA) performed | 469
  Visual Inspection with Acetic Acid (VIA) performed on the same day | 459

2. Primary Outcome: Same-day Thermocoagulation Rate Among Women Who Were HPV-positive and Ablation-eligible by Colposcopy Triage
Description: Among women who tested HPV-positive through primary screening, those eligible for thermocoagulation by colposcopy triage received thermocoagulation treatment on the same day as self-collection. As specified in the study protocol, data were not stratified by HIV status for this outcome due to lack of scientific rationale for a difference in same-day colposcopy completion by HIV status.
Time Frame: Baseline
Population: Participants who underwent HPV-based primary screening for cervical cancer and tested HPV-positive and were eligible for thermocoagulation by colposcopy triage and had thermocoagulation performed on the same day of self-collection.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Positive
Number analyzed (Participants) | 476
Participants
  HPV-positive participants eligible for thermocoagulation based on colposcopy triage | 110
  Thermocoagulation completed among HPV-positive participants on same day of self-collection | 109

3. Primary Outcome: High Risk (hr)-Human Papillomavirus (HPV) Positive Rate
Description: The proportion of women who tested High risk (hr)-human papillomavirus (HPV) positive on a self-collected vaginal brush among enrolled participants.
Time Frame: Baseline
Population: Participants joined the study and provided self-collected vaginal samples using a Viba-Brush® for HPV testing.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Positive | HIV Negative
Number analyzed (Participants) | 625 | 625
Participants | 295 | 181

4. Secondary Outcome: HPV Screen-triage-treat Algorithm for Cervical Cancer Screening
Description: To evaluate the performance of the proposed ICC screen-and-treat strategy for cervical carcinoma screening among women who are HIV- positive, the rates of overtreatment and undertreatment rates were estimated. Overtreatment for women who are HPV-positive VIA- positive/ablation-eligible and would have received thermocoagulation but had no cervical precancer (i.e., high-grade cervical intraepithelial neoplasia), and undertreatment among HPV-positive with high-grade cervical intraepithelial neoplasia but were VIA-positive and eligible for thermocoagulation, and those who were VIA-negative.
Time Frame: Up to 24 weeks
Population: Participants who tested HPV-positive for cervical cancer screening in the study and completed the screen-triage-treat algorithm.
Measure: Count of Participants; unit: Participants
Groups:
- HIV Positive, HPV Positive, VIA Positive, and Had no High Grade Cervical Intraepithelial Neoplasia: Women living with HIV, human, papillomavirus (HPV) positive, Visual Inspection with Acetic Acid test positive, and had no biopsy-proven cervical precancer but would have received thermocoagulation by VIA triage though without biopsy-proven cervical precancer.
- HIV Positive,HPV Positive, VIA Positive, and Had Biopsy-proven Cervical Precancer in the Endocervix: Women living with HIV, human, papillomavirus (HPV) positive and, Visual Inspection with Acetic Acid positive, and could have received thermocoagulation by VIA triage but had biopsy-proven cervical precancer in the endocervical epithelium (thermocoagulation might not adequately treat precancer in the endocervix.
- HIV Positive, HPV Negative, VIA Positive: Women living with HIV, human, papillomavirus (HPV) negative and Visual Inspection with Acetic Acid test positive.
Arm/Group | HIV Positive, HPV Positive, VIA Positive, and Had no High Grade Cervical Intraepithelial Neoplasia | HIV Positive,HPV Positive, VIA Positive, and Had Biopsy-proven Cervical Precancer in the Endocervix | HIV Positive, HPV Negative, VIA Positive
Number analyzed (Participants) | 74 | 42 | 38
Participants | 49 | 10 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 weeks.
Description: Adverse events were collected from day one of the study to 4 weeks after completion of the thermocoagulation intervention in participants who received thermocoagulation only. Adverse events were not monitored/assessed in any other participants.
Groups:
- HIV Positive -VIA and Thermocoagulation: HIV Positive Participants will undergo the same-day VIA and thermocoagulation were included.
- HIV Negative -VIA and Thermocoagulation: HIV HIV-negative participants will undergo the same-day VIA and thermocoagulation were included.
Arm/Group | HIV Positive -VIA and Thermocoagulation | HIV Negative -VIA and Thermocoagulation
All-Cause Mortality (participants affected / at risk) | 1/22 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/28
Other Adverse Events (participants affected / at risk) | 19/22 | 21/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV Positive -VIA and Thermocoagulation (N=22) | HIV Negative -VIA and Thermocoagulation (N=28)
Dysuria (Renal and urinary disorders) | 0 | 1
Vaginal Inflammation (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Amenorrhea (Reproductive system and breast disorders) | 0 | 2
Menorrhagia (Reproductive system and breast disorders) | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 4 | 4
vaginal bleeding (Reproductive system and breast disorders) | 1 | 4
vaginal discharge (Reproductive system and breast disorders) | 14 | 14
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 4
Hypertension (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The small sample size of women with cervical precancer and the experienced research team may limit the generalizability of findings, especially in national screening programs where providers have multiple tasks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04092257/Prot_SAP_000.pdf